CLINICAL TRIAL: NCT01629654
Title: Poststroke Fatigue - Developing and Testing a Program to Reduce and Cope With Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); The Novo Nordic Foundation (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: TEA2011
Record Dates: First submitted 2012-01-20; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Cardiovascular Disease; Stroke
Keywords: Poststroke fatigue; Health promotion; Patient education
MeSH Terms: conditions — Cardiovascular Diseases; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental): Testing of the teory- and evidence based health promotion program. Patients will participate in a 13 weeks program.
  Interventions: Behavioral: Health promotion program

INTERVENTIONS:
Behavioral: Health promotion program — A 13 weeks organized program:
  * One group session about poststroke fatigue involving both patient and relatives
  * Two personal meetings, involving both patient and relatives
  * Three telephone meetings, involving only patient
  Other Names: Poststroke fatigue; Complex interventions

SUMMARY:
Fatigue is a common complaint after stroke, reported by 39-72% of patients. Poststroke fatigue is related to poor neurological recovery, low level of activities of daily living, decreased quality of life and may possibly affect the ability to return to work. Little is known about strategies addressing post-stroke fatigue and their effectiveness.

Aim: to develop, test and evaluate a health promotion program based on strategies addressing poststroke fatigue.

DETAILED DESCRIPTION:
Fatigue is a common complaint after stroke, reported by 39-72% of patients. It has been shown that poststroke fatigue may be related to poor neurological recovery, low level of activities of daily living and decreased quality of life. However, little is known about strategies to address poststroke fatigue and the effectiveness of such strategies.

Objective The aim of the study is to develop a program based on strategies to address poststroke fatigue and to test and evaluate the program.

Material and Methods Intervention Mapping is the overall approach of the study. It describes a protocol for the development of theory- and evidence-based health promotion programmes.

Step 1) The program is developed based on a needs assessment. Existing knowledge about physical, psychosocial and environmental factors associated with poststroke fatigue is mapped in a literature review.

Step 2) The program will be tested in a pilot study (controlled trial). In addition to conventional treatment, the patients in the intervention group will participate in the program for a period of 12 weeks. The control group will receive conventional treatment only.

Step 3) Evaluation of the program: Primary outcome measure will be fatigue, measured on the Multidimensional Fatigue Inventory-20. Secondary outcome measures will be identified during the development of the program. Patients will be tested at baseline, after 3 months and after 6 months. The effect size in the pilot study will be assessed and will be used in order to estimate the required sample size for a large-scale randomized controlled trial on formally testing the efficacy of the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first ever stroke
* > 18 year
* Living in the area of Aarhus(intervention group) and patients living in the area of Holstebro (control group).
* Multidimensional Fatigue Inventory-20/Generel Fatigue > 12.
* The patient must be able to give informed consent
* Walking without person support.
* Walking aids is accepted.

Exclusion Criteria:

* Neurological problems related to acute stroke(severe aphasia, decreased level of conscience or decreased attention)
* Other neurologic or psychiatric deseases (including dementia, non treated depression, misuse of alcohol eller medicin)
* Severe co-morbidity (including cancer, blindness or deathness)
* Not-danish speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory 20 | Change from baseline in MFI-20 at 3 and 6 months
  The multidimensional Fatigue Inventory 20 is a multidimensional fatigue score covering five dimensions of fatigue: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Activity. Pathologic Fatigue is defined as a score ≥ 12 on the General Fatigue dimension.

SECONDARY OUTCOMES:
The general self-efficacy scale | Change from baseline in the generel self-efficacy scale at 3 and 6 months
  The general self-efficacy scale is a scale measuring how individuals cope with distressing situations

CONTACTS AND LOCATIONS:
Overall Officials: Marit Kirkevold, Professor, Principal Investigator — University of Aarhus, Health, Nursing Science
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus, Central Jutland, Denmark